CLINICAL TRIAL: NCT05991583
Title: A Phase I/II Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IBB0979 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Trial to Evaluate Effect of IBB0979 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IBB0979-101
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Tumors
Keywords: Advanced Malignant Tumors; B7-H3; IL-10

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia - Dose escalation (Experimental): The goal of the Dose Escalation Phase (Part A) is to initially characterize the safety and tolerability of IBB0979, and more specifically to describe the DLTs for each dose level studied and to define the MTD based on the frequency of the occurrence of DLTs in each cohort during the DLT evaluation period.
  Interventions: Drug: IBB0979
- Phase Ib - Dose extension (Experimental): During the Dose Expansion Phase , patients will be enrolled to receive IBB0979 at the MTD established from the Dose Escalation Phase of the study.
  Interventions: Drug: IBB0979
- Phase IIa - Clinical Exploratory Stage (Experimental): After finishing Phase 1, invesigators will discuss with the sponsor about how to carry out the Phase IIa due to the results acheived from Phase I.
  Interventions: Drug: IBB0979

INTERVENTIONS:
Drug: IBB0979 — IBB0979 should be subcutaneous injected，qw

SUMMARY:
This is a Phase 1/2, open-label, dose escalation and dose expansion study designed to characterize the safety, tolerability, PK, immunogenicity, and preliminary antitumor activity of IBB0979 in previously treated patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study consists of Dose Escalation Phase, Dose Expansion Phase and Clinical Exploration Phase.

Dose Escalation Phase：This phase is an open-label, non-randomized, multicenter, dose-escalation study. From the starting dose of 0.01 mg/kg, an accelerated titration combined with a "3+3" design will be adopted.

Dose Expansion Phase：The application of Dose Expansion Phase can be discussed by investigator and sponsor based on data obtained in Dose Escalation Phase. This phase is an open-label, non-randomized, multicenter study. 6 patients with locally advanced or metastatic solid tumors are expected to be enrolled at DRDE. Each treatment cycle is defined as 21 days, patient may receive treatment until withdrawal or Treatment Discontinuation.

Clinical Exploration Phase：After completing the dose escalation and expansion studies, the indication and study population can be discussed by the investigator and sponsor based on the efficacy and safety data that have been obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years old.
2. With histologically or cytologically confirmed locally advanced or metastatic solid malignant tumors, either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate.
3. There is at least one assessable tumor lesion in the Dose Escalation Phase and at least one measurable lesion in the Dose Expansion Phase According to RECIST 1.1 (tumor lesions located in the previous radiation therapy area or other local regional treatment area generally not be considered as measurable lesions, unless the lesion has progression or persists after three months of radiation therapy).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy ≥ 3 months.
6. Adequate organ functions:

   * Hematologic system (no transfusion or hematopoietic-stimulating factor therapy within 14 days): absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 90 × 109/L, hemoglobin (HGB) ≥ 90 g/L.

     * Liver function: total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal values (ULN), except for Gilbert's syndrome; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN, liver metastases or liver cancer patients with ALT and AST ≤ 5.0 × ULN.

       * Renal function: estimated creatinine clearance (Ccr) ≥ 50 mL/min (calculated according to the Cockcroft-Gault formula).

         * Thrombin function: international normalized ratio of prothrombin (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
7. Eligible patients with fertility (male and female) must agree to use reliable contraceptive measures (include hormonal contraceptives, barrier contraception or abstinence) with their partners from the time of consent through 90 days after discontinuation of investigational product administration. Female patients of childbearing potential (not surgically sterilized and between menarche and 1- year postmenopause) must have a negative serum pregnancy test within 7 days prior to the initiation of investigational product administration.
8. Ability to provide informed consent and documentation of informed consent prior to initiation of any study-related tests or procedures.

Exclusion Criteria:

1. Known hypersensitivity (≥ Grade 3) to recombinant proteins or any excipient contained in the drug or vehicle formulation for IBB0979.
2. History of anti-tumor therapy (chemotherapy within 3 weeks or radiotherapy, biological therapy, endocrine therapy, targeted therapy within 4 weeks) prior to the initiation of investigational product administration, with the following exceptions:

   * Nitrosourea or mitomycin C should be within 6 weeks prior to the initiation of investigational product administration.

     * Oral fluoropyrimidines and small molecule targeted drugs should be within 2 weeks prior to the initiation of investigational product administration.
3. History of any un-marketed investigational product or therapy within 4 weeks prior to the initiation of investigational product administration.
4. History of major organ surgery (with exception of aspiration biopsy) or significant trauma within 4 weeks prior to the initiation of investigational product administration, or selective operation is required during the trial.
5. History of systemic corticosteroids (prednisone >10 mg per day or equivalent) or other immune-suppressive drugs within the 14 days prior to the initiation of investigational product administration. Steroids for topical, ophthalmic, intraarticular, inhaled or nasal administration are allowed.
6. Treatment with immunomodulatory agents, including but not limited to thymosin, interleukin-2 and interferon within 14 days prior to the initiation of investigational product administration.
7. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of investigational product administration.
8. History of prior allogeneic stem-cell or solid organ transplantation.
9. The adverse effects of previous anti-tumor therapy have not yet returned to ≤ Grade 1 (NCI-CTCAE 5.0) or rules of the inclusion criteria (with exception of that the investigator judged to be without safety risks, such as hair loss, Grade 2 peripheral neurotoxicity, stable hypothyroidism with hormone replacement therapy, etc.).
10. Active brain or leptomeningeal metastases with clinical symptoms. Patients with brain metastases are eligible if these have been treated and MRI or CT shows no evidence of progression for at least 8 weeks after treatment completion and within 4 weeks prior to the initiation of investigational product.
11. Evidence of active infection requiring intravenous anti-infective therapy.
12. Active hepatitis B (HBsAg-positive, and HBV-DNA> 500 IU/mL or lower limit of study site [only if the lower limit of study site is above 500 IU/mL]), active hepatitis C (HCV-RNA> lower limit of study site).
13. Currently has interstitial lung disease (with exception of radiation pulmonary fibrosis that requires no hormone therapy).
14. History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    * Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II/III-degree atrioventricular block, etc.

      * The mean QT interval (QTcF) > 470 ms corrected by Fridericia's method.

        * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of ≥ grade 3 within 6 months prior to the initiation of investigational product.

          * Congestive heart failure (New York Heart Association [NYHA] class ≥ grade II) or left ventricle ejection fraction (LVEF) < 50%, or other structural heart disease at high risk by the investigator.

            * Clinically uncontrolled hypertension.
15. Active or suspected autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), with exception of clinically stable autoimmune thyroid disease, type I diabetes, vitiligo, cured atopic dermatitis in children and psoriasis without systemic treatment (within the past 2 years).
16. History of ≥ grade 3 immune-related adverse events (irAE) or Grade 2 immune-associated myocarditis accompanied with immunotherapy, with exception of ≥ Grade 3 immune-associated thyrotoxicosis.
17. History of another malignancy or a concurrent malignancy. Exceptions include patients who have been disease free for two years for non-melanoma skin cancer, localized prostate cancer or carcinoma in situ (e.g., cervical cancer in situ), etc.
18. Clinically uncontrolled effusion in the third space, which is unsuitable for participation in the study by the investigator.
19. Known alcohol or drug dependence.
20. History of mental disorder or poor adherence.
21. The female patient who is pregnant or breastfeeding. History of other severe systemic disease, or any issue that in the opinion of the investigator, would contraindicate the patient's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Dose limiting toxicities (DLTs) (Phase Ⅰ) | 21 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
Objective response rate (ORR) in dose expansion (Phase Ⅱa) | Baseline through up to 1 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmax) following single dose.following single dose.
Pharmacokinetic (PK) Cmin (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmin) following single dose.following single dose.
Pharmacokinetic (PK) Tmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-t) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) CL (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CL) following single dose.
Pharmacokinetic (PK) Vd (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vd) following single dose.
Pharmacokinetic (PK) t1/2 (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,max) following multiple dose.
Pharmacokinetic (PK) Css,min (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,min) following multiple dose.
Pharmacokinetic (PK) Css,av (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,av) following multiple dose.
Pharmacokinetic (PK) AUCss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUCss) following multiple dose.
Pharmacokinetic (PK) CLss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CLss) following multiple dose.
Pharmacokinetic (PK) Vss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vss) following multiple dose.
Pharmacokinetic (PK) R (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (R) following multiple dose.
Pharmacokinetic (PK) DF (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (DF) following multiple dose.
Objective response rate (ORR) in dose escalation (Phase Ⅰ) | Baseline through up to 1 years or until disease progression
  Tumor response based on RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IBB0979 | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IBB0979.(Phase Ⅰb)
Progression free survival (PFS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1.
Overall survival (OS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
Disease control rate (DCR) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  To investigate the safety characteristics.
Immunogenicity of IBB0979 (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  The frequency of anti-drug antibodies (ADA) against IBB09798.(Phase Ⅱa)

CONTACTS AND LOCATIONS:
Overall Officials: Li Jin, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China